CLINICAL TRIAL: NCT05343975
Title: Evaluating the Value of Audio-guided Meditation During Breast Biopsy Procedures
Acronym: MAG-BM
Status: Completed | Type: Observational
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Other Study IDs: ICO-2021-31
Record Dates: First submitted 2022-03-11; First posted 2022-04-25 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-08

CONDITIONS: Breast Disease
MeSH Terms: conditions — Breast Diseases | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: biopsy with audio-guided Meditation — biopsy with audio-guided Meditation

SUMMARY:
A prospective, non-randomized, single-center cohort study to evaluate the value of audio-guided meditation during breast biopsy procedures.

The main criterion of judgment is based on the evaluation of tolerance, which includes anxiety and pain felt. This is assessed with questionnaires (STAI-ETAT and EN) before and after the procedure.

Secondary endpoints include tolerance of additional physical pain, reduction in the number of per-procedure complications, overall satisfaction of the practitioner with the biopsy procedure, and comparison of the tolerance of the procedure in patients who practice meditation at home before the procedure

DETAILED DESCRIPTION:
audio-guided meditation during breast biopsy procedures questionnaires (STAI-ETAT and EN) before and after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Breast pathology requiring the performance of one (or more) breast and/or axillary micro or macrobiopsy,
* Informed patient, with collection of the non opposition

Exclusion Criteria:

* Excluded forms of the disease: biopsy concerning organs other than the breast and/or axilla
* Persons deprived of their liberty, under court protection, under curatorship or under the authority of a guardian,
* Impossibility to submit to the medical follow-up of the trial for geographical, social or psychic reasons (invalidating psychiatric disorder diagnosed of psychotic type).

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women referred to the ICO of Angers for management of a breast pathology, or during screening, requiring the performance of one (or more) breast micro or macrobiopsy.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
To describe the level of pain according to whether or not patients listen to audio-guided mediation during the breast biopsy procedure | immediately after procedure
  11-point numerical scale (from 0 = no pain to 10 = maximal pain)
To describe anxiety according to whether or not patients listen to audio-guided mediation during the breast biopsy procedure | immediately after procedure
  State Trait Anxiety Inventory Etat - Trait (40 questions - each item has a score from 1 to 4 (4 being the highest level of anxiety))

SECONDARY OUTCOMES:
per-biopsy complications | immediately after procedure (same day of the biopsy)
  complications
satisfaction of the radiologist with regard to the procedure | immediately after procedure
  questions about 1. overall quality of the doctor-patient relationship and 2. Patient compliance with the procedure with scales in 4 point
efficacy of the procedure | immediately after procedure
  number of samples taken in the target

CONTACTS AND LOCATIONS:
Overall Officials: Pierre BERGE, MD, Principal Investigator — INSTITUT DE CANCEROLOGIE DE L'OUEST
Locations (1):
- Institut de Cancerologie de L'Ouest (Ico), Angers, France

IPD SHARING:
Plan to Share IPD: No